CLINICAL TRIAL: NCT02877095
Title: Subcutaneous Furosemide in Acute Decompensated Heart Failure: The SUBQ-HF Pilot Study
Brief Title: Subcutaneous Furosemide in Acute Decompensated Heart Failure Pilot
Acronym: SUBQ-Pilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adrian Hernandez (Other)
Responsible Party: Sponsor-Investigator, Adrian Hernandez, HFN Coordinating Center PI, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00070399
Record Dates: First submitted 2016-08-15; First posted 2016-08-24 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active (Experimental): All subjects in the pilot study will receive the subcutaneous pump to administer a special formulation of furosemide to be delivered subcutaneously.
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — subcutaneous furosemide delivered via subcutaneous pump
  Other Names: Lasix

SUMMARY:
The Pilot study is designed to evaluate the overall safety and feasibility of a strategy based on subcutaneous delivery of furosemide. It will be used to inform the subsequent evaluation phase of the study (separate protocol). The primary objective of the study is to determine if a strategy of a novel subcutaneous delivery of furosemide is safe and feasible in patients with acute heart failure.

DETAILED DESCRIPTION:
Multi-center, open-label, pilot study conducted in 2 phases. Each phase will enroll 20 subjects that will be used to inform the study design of the SUBQ-HF Study (approximately 300 evaluable patients randomized to either usual inpatient care or early discharge with home subcutaneous furosemide for 1-7 days).

Inpatient Pilot Phase:

Eligible in-patients will be approached for participation. Subjects who consent for participation will be treated with subcutaneous furosemide for 48 hours, during which they will remain in the hospital. This will be primarily a safety and feasibility assessment. There will be no formal hypothesis tested, and statistical analysis will be descriptive in nature.

Outpatient Pilot Phase:

Eligible in-patients who are nearing discharge will be approached for participation. Subjects who consent for participation will be instructed on use of device, discharged to home and treated at home with subcutaneous furosemide for 1-7 days. This will be primarily a safety and feasibility assessment. There will be no formal hypothesis tested, and statistical analysis will be descriptive in nature.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Willingness and ability to provide informed consent
3. Hospitalization for acute heart failure (AHF) with at least 1 symptom (dyspnea, orthopnea, or edema) AND 1 sign (rales on auscultation, peripheral edema, ascites, pulmonary vascular congestion on chest radiography, Brain Natriuretic Peptide > 250 ng/mL or N-terminal pro-brain natriuretic peptide (NTproBNP) > 1000 ng/mL) of congestion
4. Persistent congestion despite at least 18 hours of intravenous (IV) therapy, defined by the presence of at least 2 or more of the following at the time of consent:

   * Peripheral edema
   * Rales
   * Elevated jugular venous pressure (JVP)
   * Ascites
   * BNP > 250 ng/mL or NTproBNP > 1000 ng/mL
5. Total anticipated daily IV furosemide dose (at time of screening) >80-200 mg (or equivalent)/day
6. Anticipated need for at least 24 more hours of parenteral diuretic therapy -

Exclusion Criteria:

1. Severe renal dysfunction (Estimated Glomerular Filtration Rate (eGFR)< 30 ml/min/1.73m2)
2. Requirement for inotropes (other than digoxin) or mechanical support during hospitalization
3. Clinically significant electrical instability during hospitalization
4. Ongoing need for other intravenous therapies beyond diuretics (vasodilators, antibiotics, etc.)
5. Anticipated need for ongoing parenteral electrolyte repletion
6. Planned discharge to location other than home (e.g, hospice, skilled nursing facility, etc.)
7. Anticipated cardiac transplantation or left ventricular assist device within the next 30 days
8. Primary hypertrophic cardiomyopathy, infiltrative cardiomyopathy, acute myocarditis, constrictive pericarditis or tamponade
9. Known or anticipated pregnancy in the next 30 days Prior use of subcutaneous furosemide pump or current use of any subcutaneous pump, on-body infusion devices or patients who give regimented injections at the intended site of the furosemide infusion device
10. Other psychosocial or physical barriers to following the protocol and using a subcutaneous pump device outside the hospital setting
11. Unable to accurately measure urine output
12. Known allergy to furosemide
13. Known sensitivity or allergy to medical adhesive tape

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD, Principal Investigator — Duke University; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (5):
- United States (5):
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Metro Health System, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- In-patient Pilot: All subjects in the in-patient study will receive the subcutaneous pump to administer a special formulation of furosemide to be delivered subcutaneously.
  Furosemide: subcutaneous furosemide delivered via subcutaneous pump
- Out-patient Pilot Study: All subjects in the out-patient study will receive the subcutaneous pump to administer a special formulation of furosemide to be delivered subcutaneously.
  Furosemide: subcutaneous furosemide delivered via subcutaneous pump
Period: Overall Study
Arm/Group | In-patient Pilot | Out-patient Pilot Study
Started | 20 (First patient enrolled 1/9/17.) | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- In-patient Pilot Study: All subjects in the in-patient pilot study will receive the subcutaneous pump to administer a special formulation of furosemide to be delivered subcutaneously.
  Furosemide: subcutaneous furosemide delivered via subcutaneous pump
- Total: Total of all reporting groups
Arm/Group | In-patient Pilot Study | Out-patient Pilot Study | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (14.6) | 57.8 (12.0) | 63.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 12 | 16 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety of a Strategy Based on Subcutaneous Delivery of Furosemide in Inpatients and Outpatients as Measured by Number of Adverse Events
Description: The analysis of data from the Pilot Phase will be primarily descriptive in nature and there will be no formal hypothesis testing. Number of patients with events will be reported.
Time Frame: 14 days
Measure: Number; unit: participants
Groups:
- In-patient Pilot; Out-patient Pilot Study: All subjects in the pilot study will receive the subcutaneous pump to administer a special formulation of furosemide to be delivered subcutaneously.
  Furosemide: subcutaneous furosemide delivered via subcutaneous pump
Arm/Group | In-patient Pilot | Out-patient Pilot Study
Number analyzed (Participants) | 20 | 20
participants
  Patients with any Adverse Events | 4 | 9
  Patients with no Events | 16 | 11
Statistical Analysis 1: Comparison: In-patient Pilot; All subjects on study received active drug; Test type: Other; Total count of events is provided

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- In-patient Pilot Study: All subjects in the in-patient study will receive the subcutaneous pump to administer a special formulation of furosemide to be delivered subcutaneously.
  Furosemide: subcutaneous furosemide delivered via subcutaneous pump
Arm/Group | In-patient Pilot Study | Out-patient Pilot Study
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 4/20 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-patient Pilot Study (N=20) | Out-patient Pilot Study (N=20)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | In-patient Pilot Study (N=20) | Out-patient Pilot Study (N=20)
Injection Site Pain (General disorders) | 2 (2) | 2 (2)
Injection Site discomfort (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site haemorhage (General disorders) | 0 (0) | 1 (1)
Injection Site Rash (General disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT02877095/Prot_SAP_000.pdf